CLINICAL TRIAL: NCT02991430
Title: A Non-Invasive Neuromodulation Device for Prevention of Episodic Migraine Headache
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to supply and maintain treatment device. No safety concerns occurred.
Sponsor: Scion NeuroStim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SNS-MIG-02
Record Dates: First submitted 2016-12-04; First posted 2016-12-13 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Intervention
Keywords: migraine headache, episodic
MeSH Terms: conditions — Migraine Disorders; Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- active (Active Comparator): active neuromodulation
  Interventions: Device: active neuromodulation for episodic migraine headache
- placebo (Placebo Comparator): placebo neuromodulation
  Interventions: Device: placebo neuromodulation for episodic migraine headache

INTERVENTIONS:
Device: active neuromodulation for episodic migraine headache — Non-invasive brainstem neuromodulator. Active and placebo devices appear identical
  Arms: active
Device: placebo neuromodulation for episodic migraine headache — Sham non-invasive brainstem neuromodulator. Active and placebo devices appear identical
  Arms: placebo

SUMMARY:
This study will assess the efficacy of a neuromodulation device for the treatment of episodic migraine headache.

DETAILED DESCRIPTION:
This study is a multi-center, triple-blinded, placebo-controlled, randomized clinical trial for adjunctive prophylactic treatment of episodic migraine headache (with or without aura) using neuromodulation device developed by Scion NeuroStim, LLC (SNS). The investigational use of the device for episodic migraine headache has been reviewed by the FDA and is classified as NSR (non-significant risk).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with episodic migraine at least 6 months before study
* at least 3 consecutive months of stable migraine headaches before study
* at least 4-14 headache days per month, of which 4-14 may be migraines
* must not have failed on more than 2 classes of migraine preventatives

Exclusion Criteria:

* previous use of the experimental device
* pregnant
* using more than 1 concurrent migraine preventive
* history of cardiovascular disease
* work night shifts
* diagnosed with vestibular migraine
* menstrual migraines exclusively
* diagnosed with post-traumatic migraine
* have a history of unstable mood or anxiety disorder
* use a hearing aid
* have a cochlear implant
* have chronic tinnitus
* have temporomandibular joint disease
* diagnosed with traumatic brain injury
* diagnosed with neurological disease other than headaches
* diagnosed vestibular and/or balance dysfunction
* history of abusing alcohol or other drugs
* are experiencing medication overuse headaches
* have had eye surgery in the previous 3 months
* have had ear surgery in the previous 6 months
* have active ear infections or a perforated tympanic membrane
* have participated in another clinical trial in the last 30 days
* are currently participating in another clinical trial
* using Botulinum toxin-based treatments for migraines or cosmetic reasons
* taking anti-emetics more than 2 times per week (consistently)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (8):
  - Mayo Clinic, Scottsdale, Arizona
  - Neurology Research Institute, West Palm Beach, Florida
  - Diamond Headache Clinic, Chicago, Illinois
  - Michigan Headache Pain & Neurological Inst., Ann Arbor, Michigan
  - Study Metrix Research, City of Saint Peters, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cleveland Clinic, Cleveland, Ohio
  - Jefferson Headache Center, Philadelphia, Pennsylvania
- United Kingdom (2):
  - King's College London, London, Denmark Hill
  - University of Kent, Canterbury, Kent

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BID Placebo: Participants self-administered twice-daily inactive/sham treatments for 12 weeks (treatment period 1) followed by twice-daily active treatments for 12 weeks (treatment period 2) followed by a post-treatment observation period lasting 12 weeks (observation period).
- BID Active: Participants self-administered twice-daily active treatments for 12 weeks (treatment period 1) followed by twice-daily active treatments for an additional 12 weeks (treatment period 2) followed by a post-treatment observation period lasting 12 weeks (observation period).
- QD Active: Participants self-administered once-daily active treatments for 12 weeks (treatment period 1) followed by once-daily active treatments for an additional 12 weeks (treatment period 2) followed by a post-treatment observation period lasting 12 weeks (observation period).
Period: Treatment Period 1
Arm/Group | BID Placebo | BID Active | QD Active
Started | 14 | 15 | 16
Completed | 13 | 11 | 14
Not Completed | 1 | 4 | 2
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 4 | 0
Period: Treatment Period 2
Arm/Group | BID Placebo | BID Active | QD Active
Started | 13 | 11 | 14
Completed | 7 | 8 | 10
Not Completed | 6 | 3 | 4
Not completed — Study Termination | 6 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Period: Post-treatment Observation Period
Arm/Group | BID Placebo | BID Active | QD Active
Started | 7 | 8 | 10
Completed | 4 | 2 | 5
Not Completed | 3 | 6 | 5
Not completed — Study Termination | 3 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- BID Placebo: Participants self-administered twice-daily inactive/sham treatments for 12 weeks followed by twice-daily active treatments for 12 weeks followed by a post-treatment observation period lasting 12 months.
- BID Active: Participants self-administered twice-daily treatments for 12 weeks followed by twice-daily active treatments for an additional 12 weeks followed by a post-treatment observation period lasting 12 months.
- QD Active: Participants self-administered once-daily treatments for 12 weeks followed by once-daily active treatments for an additional 12 weeks followed by a post-treatment observation period lasting 12 months.
- Total: Total of all reporting groups
Arm/Group | BID Placebo | BID Active | QD Active | Total
Number analyzed (Participants) | 14 | 15 | 16 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (12.2) | 43.9 (11.3) | 43.5 (10.8) | 43.87 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 14 | 37
  Male | 2 | 4 | 2 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Monthly migraine days [Mean (Standard Deviation); unit: days] — Monthly migraine days within the 28 day baseline according to an electronic daily diary.
  days | 7.9 (1.7) | 7.7 (1.9) | 7.5 (2.4) | 7.8 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Migraine Headache Days (MHD)
Description: comparison of MHD recorded in baseline month versus 3rd month of treatment
Time Frame: 1 month of baseline recordation followed by 84 days of device use
Population: The majority of devices failed in the field, preferentially affecting the active arm/group. As a result, data collection was compromised due to the frequent device failures and thus the results are not reported. No significant device related AE's were reported over the course of the Study.
Arm/Group | BID Placebo | BID Active | QD Active
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Normalized Reduction in Migraine Headache Days
Description: comparison of MHD recorded in baseline month versus 3rd month of treatment: percentages, active versus placebo
Time Frame: 1 month of baseline recordation followed by 84 days of device use
Population: as for outcome 1
Arm/Group | BID Placebo | BID Active | QD Active
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change in Medication Usage
Description: reduction in acute, prescribed medications in month 3 of treatment versus baseline month
Time Frame: 1 month of baseline recordation followed by 84 days of device use
Population: as for outcome 1
Arm/Group | BID Placebo | BID Active | QD Active
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change in Headache Pain
Description: reduction in subject perceived headache pain scores in month 3 of treatment versus baseline month
Time Frame: 1 month of baseline recordation followed by 84 days of device use
Population: as for outcome 1
Arm/Group | BID Placebo | BID Active | QD Active
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change in Quality of Life
Description: comparison of HIT-6 (headache impact test) scores between baseline month and treatment month 3
Time Frame: 1 month of baseline recordation followed by 84 days of device use
Population: as for outcome 1
Arm/Group | BID Placebo | BID Active | QD Active
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change in Depression
Description: comparison of BDI-II (Beck depression index) scores between baseline month and treatment month 3
Time Frame: 1 month of baseline recordation followed by 84 days of device use
Population: as for outcome 1
Arm/Group | BID Placebo | BID Active | QD Active
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Change in Anxiety
Description: comparison of BAI (Beck anxiety index) scores between baseline month and treatment month 3
Time Frame: 1 month of baseline recordation followed by 84 days of device use
Population: as for outcome 1
Arm/Group | BID Placebo | BID Active | QD Active
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change in Sleep Quality
Description: comparison of Pittsburgh Sleep assessment scores between baseline month and treatment month 3
Time Frame: 1 month of baseline recordation followed by 84 days of device use
Population: as for outcome 1
Arm/Group | BID Placebo | BID Active | QD Active
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Additional Treatment Time
Description: comparison of MHD recorded in baseline month versus 6th month of treatment
Time Frame: 1 month of baseline recordation followed by 168 days of device use
Population: as for outcome 1
Arm/Group | BID Placebo | BID Active | QD Active
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Sustained Reduction in Migraine Headache Days
Description: comparison of MHD recorded in baseline month versus post-treatment months 7, 8 and 9
Time Frame: 1 month of baseline recordation followed by 252 days of device use
Population: as for outcome 1
Arm/Group | BID Placebo | BID Active | QD Active
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | BID Placebo | BID Active | QD Active
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 4/14 | 7/15 | 4/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BID Placebo (N=14) | BID Active (N=15) | QD Active (N=16)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 1 (2)
Ear discomfort, itch, irritation, pruritis or fullness (Product Issues) | 3 (3) | 7 (9) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT02991430/Prot_SAP_000.pdf